CLINICAL TRIAL: NCT02787980
Title: Dosage of Serum Tryptase Levels in a Population of Premature Newborns to Evaluate Mast Cell Activity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: PO14087
Record Dates: First submitted 2016-05-12; First posted 2016-06-02 (Estimated); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Premature Newborns

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Patients = premature newborns (Other): "Patients" will consist of all premature babies (<37 weeks of amenorrhea), managed in the first 24 hours of life at the Reims university hospital for whom parents accepted to participate in the research Additional taking blood
  Interventions: Biological: Additional taking blood
- "Controls" = children born full term (Other): For "controls" the participation to research would be proposed to parents of children born full term, just after each "patient" child included.
  Additional taking blood
  Interventions: Biological: Additional taking blood

INTERVENTIONS:
Biological: Additional taking blood — Additional blood collection of 1 ml during the biological workup usually done.

SUMMARY:
Compare serum tryptase levels of premature babies (<37 weeks of amenorrhea) to children born at full term.

Study the evolution of serum tryptase levels in premature babies(<37 weeks of amenorrhea). Study the relationship between the onset of infectious complications, mainly the type of necrotizing enterocolitis seen in premature babies (<37 weeks of amenorrhea) and the evolution profile of serum tryptase levels.

DETAILED DESCRIPTION:
It seems appropriate to believe that prematurity associated or not with a genetic-related sensitivity, involving several signaling pathways, makes children more vulnerable to different environmental, infectious factors that could trigger the different pathologies of premature babies. Mast cell, via its mediators, seems to play a key role.

Dosage of serum tryptase levels which is easily accessible and the work by Vitte let us imagine that the younger the child, the greater the mast cell expression, thus opening a capital pathway in the comprehension of immune system phenomena in premature babies and investigators can hope that by performing regular workups of serum tryptase levels, investigators could validate that some premature babies will express this activity in a more important manner. The relationship to eventual pathological phenomena such as necrotizing enterocolitis, but also bronchopulmonary dysplasia could then be highlighted.

ELIGIBILITY:
Inclusion Criteria "Patients" :

* all premature babies (<37 weeks of amenorrhea)
* managed in the first 24 hours of life at the Reims university hospital
* parents accepted to participate in the research - social security card

Inclusion Criteria "Controls" :

* children born full term, just after each "patient" child included
* managed in the first 24 hours of life at the Reims university hospital
* parents accepted to participate in the research.

Exclusion Criteria "Patients" and "Controls"

* Not managed in the first 24 hours of life at the Reims University Hospital,
* Person, who has parental authority, protected by law,
* Newborns with a life and death emergency in the first 24 h of life,
* Person, who has parental authority, under age 18

Max Age: 1 Month | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 87 (Actual)
Dates: Start 2015-10-12 (Actual); Primary Completion 2018-06-05 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
serum tryptase levels | infants born before 37 weeks of gestation:Day 1, day 7 and then every 15 days until new borns go home(up to 4 months). infants born after 37 weeks of gestation at Day 3

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Reims, Reims, France